CLINICAL TRIAL: NCT01492374
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and the Effect of BMS-241027 on Cerebrospinal Fluid Biomarkers in Subjects With Mild Alzheimer's Disease
Brief Title: Study to Evaluate the Safety, Tolerability and the Effect of BMS-241027 on Cerebrospinal Fluid Biomarkers in Subjects With Mild Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN167-003; 2011-004065-33 (EudraCT Number)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2013-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: BMS-241027 (0.003 mg/kg) (Experimental)
  Interventions: Drug: BMS-241027
- Arm 2: BMS-241027 (0.01 mg/kg) (Experimental)
  Interventions: Drug: BMS-241027
- Arm 3: BMS-241027 (0.03 mg/kg) (Experimental)
  Interventions: Drug: BMS-241027
- Arm 4: Placebo matching BMS-241027 (Experimental)
  Interventions: Drug: Placebo matching BMS-241027

INTERVENTIONS:
Drug: BMS-241027 — Intravenous (IV), 0.003 mg/kg, Once Weekly, 9 weeks
  Arms: Arm 1: BMS-241027 (0.003 mg/kg)
Drug: BMS-241027 — Intravenous (IV), 0.01 mg/kg, Once Weekly, 9 weeks
  Arms: Arm 2: BMS-241027 (0.01 mg/kg)
Drug: BMS-241027 — Intravenous (IV), 0.03 mg/kg, Once Weekly, 9 weeks
  Arms: Arm 3: BMS-241027 (0.03 mg/kg)
Drug: Placebo matching BMS-241027 — Intravenous (IV), 0.0 mg/kg, Once Weekly, 9 weeks
  Arms: Arm 4: Placebo matching BMS-241027

SUMMARY:
The purpose of the study is to evaluate safety and the pharmacodynamic effects of BMS-241027 on cerebrospinal fluid (CSF) Tau, connectivity magnetic resonance imaging (MRI), and computerized cognitive tests in mild Alzheimer's disease (AD) subjects, following 9 weekly intravenous (IV) infusions of BMS-241027

ELIGIBILITY:
Inclusion Criteria:

* Mild AD Subjects meeting National Institute of Neurological Disorders and Stroke - Alzheimer's Disease Related Disorders Association(NINCDS-ADRDA) and Diagnostic and Statistical Manual of Mental Disorders-Forth Edition, Text Revision (DSM-IV-TR) criteria
* Mini-Mental State Exam (MMSE) Score between 20 & 26 (inclusive)
* CSF consistent with AD pathology
* Screening brain MRI - normal - commensurate with age or demonstrate atrophy consistent with AD diagnosis (dx); reveal no more than mild white matter disease; up to 2 lacunar infarcts acceptable except in anterior thalamus, genu of internal capsule or basal forebrain; reveal no cortical infarcts; reveal no more than 4 microbleeds; reveal no focal asymmetric lobar atrophy or other findings suggesting primary cause of dementia is attributed to a cause other than AD; reveal no macrohemorrhages (>10 mm)
* Subjects must have reliable study partners
* Men and Women of Non Child Bearing Potentia (WONCBP), ages 50-90 years

Exclusion Criteria:

* Subjects with any other medical condition other than mild AD that could explain subjects' memory or cognitive deficits
* Subjects diagnosed with moderate or severe AD per DSM-IV criteria
* Subjects with a history (hx) of stroke
* Subjects with a hx of GI illnesses
* Subjects with Vitamin B12 or folate deficiency
* Subjects with any unstable cardiovascular (CV), pulmonary, Gastrointestinal (GI) or hepatic disease within 30 days prior to screening
* Subjects with active liver dx or history of hepatic intolerance
* Subjects with a Geriatric Depression Scale score of ≥ 6 at screening
* Subjects treated for or have had a diagnosis of schizophrenia
* Subjects treated for or have had a diagnosis of bipolar disease within 3 years prior to screening
* Subjects with a history of generalized peripheral neuropathy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety assessments: based on frequency of Serious Adverse Events (SAEs), frequency of Adverse events (AEs), discontinuation due to AEs and dose reduction | Within the first 70 day after first dose
Biomarker Measures: CSF levels of Tau N-terminal domain fragments | Within the first 70 day after first dose

SECONDARY OUTCOMES:
Effects of BMS-241027 on CSF levels of the mid-domain Tau fragment | Within the first 70 days after first dose
Effects of BMS-241027 on cognitive performance using computerized cognitive tests | Weeks 3, 6 and 9
Effects of BMS-241027 on connectivity MRI | Within the first 70 days after first dose
Maximal observed plasma concentration (Cmax) of BMS-241027 in subjects with mild Alzheimer's disease | Weeks 1, 4, and 9
  Intensive pharmacokinetic parameter Cmax will be derived from subgroups of subjects at Week 7
Observed plasma concentration at 24 hours post dose (C24) of BMS-241027 in subjects with mild Alzheimer's disease | Weeks 1, 4, and 9
  Intensive pharmacokinetic parameter C24 will be derived from subgroups of subjects at Week 7
Time of maximal observed plasma concentration (Tmax) of BMS-241027 in subjects with mild Alzheimer's disease | Weeks 1, 4, and 9
  Intensive pharmacokinetic parameter Tmax will be derived from subgroups of subjects at Week 7
Area under the concentration-time curve in one dosing interval [AUC(TAU)] of BMS-241027 in subjects with mild Alzheimer's disease | Weeks 1, 4, and 9
  Intensive pharmacokinetic parameter AUC(TAU) will be derived from subgroups of subjects at Week 7
Safety assessments: based on vital sign measurements, ECGs and clinical laboratory tests | Within the first 70 day after first dose
Effects of BMS-241027 on CSF levels of neurofilaments | Within the first 70 days after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (15):
  - Anaheim Clinical Trials Llc, Anaheim, California
  - Long Beach, California
  - Ucsf Memory And Aging Center, San Francisco, California
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Associated Neurologists Of Southern Connecticut, P.C., Fairfield, Connecticut
  - Compass Research, Llc, Orlando, Florida
  - Palm Beach Neurological Center Advanced Research Consultants, Palm Beach Gardens, Florida
  - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Brigham And Women'S Hospital, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - The Ohio State University, Columbus, Ohio
  - The Clinical Trial Center, Llc, Jenkintown, Pennsylvania
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Memory Center, Philadelphia, Pennsylvania
  - Lifetree Clinical Research, Salt Lake City, Utah
- Canada (3):
  - Local Institution, London, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Greenfield Park, Quebec
- France (3):
  - Local Institution, Toulouse, Cedex 9
  - Local Institution, Lille
  - Local Institution, Paris
- Germany (2):
  - Local Institution, Berlin
  - Local Institution, Heidelberg
- Local Institution, Stockholm, Sweden

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx